CLINICAL TRIAL: NCT00971802
Title: A Phase 1, Double-Blind (Sponsor Open), Randomized, Placebo- Controlled, Parallel Group, Oral Multiple-Dose Trial to Evaluate The Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PF-03882845 in Healthy Volunteers
Brief Title: A Study To Evaluate The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of PF-03882845 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: B0171008
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — (3S,3aR)-2-(3-chloro-4-cyanophenyl)-3-cyclopentyl-3,3a,4,5-tetrahydro-2H-benzo(g)indazole-7-carboxylic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): Healthy volunteers - PF-03882845 versus Placebo
  Interventions: Drug: PF-03882845 or Placebo
- Cohort 2 (Experimental): Healthy volunteers - PF-03882845 versus Placebo
  Interventions: Drug: PF-03882845 or Placebo
- Cohort 3 (Experimental): Healthy volunteers - PF-03882845 versus Placebo
  Interventions: Drug: PF-03882845 or Placebo
- Cohort 4 (Experimental): Healthy volunteers - PF-03882845 versus Placebo
  Interventions: Drug: PF-03882845 or Placebo

INTERVENTIONS:
Drug: PF-03882845 or Placebo — PF-03882845 20 mg or Placebo, daily for 10 days.
  Arms: Cohort 1
Drug: PF-03882845 or Placebo — PF-03882845 60 mg or Placebo, daily for 10 days.
  Arms: Cohort 2
Drug: PF-03882845 or Placebo — PF-03882845 120 mg or Placebo, daily for 10 days.
  Arms: Cohort 3
Drug: PF-03882845 or Placebo — PF-03882845 185 mg or Placebo, daily for 10 days.
  Arms: Cohort 4

SUMMARY:
To evaluate the safety and tolerability of PF-03882845 in Healthy Volunteers. To evaluate the pharmacokinetics of PF-03882845 in Healthy Volunteers. To evaluate the pharmacodynamics of PF-03882845 in Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant disease.
* Past medical history of epididymitis, orchitis, sexually transmitted diseases (chlamydia, gonorrhea, etc.) or urinary tract infection.
* History of prostatitis or prostate surgery.
* Urinary catheterization or instrumentation within 12 months of screening. Inguinal or scrotal hernia.
* Current or history of congenital genital abnormalities.
* Baseline scrotal ultrasound scan showing unilateral or bilateral scrotal blood flow abnormalities or anatomic abnormalities (hydrocele, cysts, other), with the exception of small epididymal cysts and spermatoceles.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing.
* History of sensitivity to spironolactone, eplerenone, or related compounds.
* Serum potassium >5.5 mEq/L at screening or Day 0.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Single-Dose PK for PF-03382845: Cmax(ss), Tmax(ss), AUC(tau,ss), half life, Cmin(ss), Cave(ss), Ae%, CL/F, V/F, CL renal; accumulation ratios AUC(tau,ss)/AUC(tau,sd) and Cmax(ss)/Cmax(sd) | 13 days
Safety and tolerability of PF-03382845 as determined by adverse event reporting, clinical laboratory results, vital signs (supine blood pressure and heart rate), physical examinations, electrocardiograms (ECGs) and potential sex hormone mediators. | 13 days

SECONDARY OUTCOMES:
Area under the effect curve (AUEC) for serum aldosterone and PRA on Day 0 and on Days 1 and 10 after administration of PF-03882845 | 11 days
Change from baseline(Day 0) to Day8 in exploratory mRNA gene expression biomarkers (SGK1:Sodium-and Serum/glucocorticoid regulated kinase 1 gene,ENaCα:Epithelial Sodium Channel alpha subunit,ENaCγ:Epithelial Sodium Channel gamma | 9 days
subunit,MR: Mineral corticoid Receptor,ACTβ:Beta Actin) after administration of PF-03882845 or placebo.These results will not be included in the study report | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, South Miami, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0171008&StudyName=A%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%2C%20And%20Pharmacodynamics%20Of%20PF-03882845%20In%20Healthy%20Volunteers